CLINICAL TRIAL: NCT04348695
Title: Randomized Phase II Clinical Trial of Ruxolitinib Plus Simvastatin in the Prevention and Treatment of Respiratory Failure of COVID-19.Ruxo-Sim-20 Clinical Trial.
Brief Title: Study of Ruxolitinib Plus Simvastatin in the Prevention and Treatment of Respiratory Failure of COVID-19.
Acronym: Ruxo-Sim-20
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación de investigación HM (Other)
Collaborators: Apices Soluciones S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ruxo-Sim-20; 2020-001405-23 (EudraCT Number)
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Coronavirus Infection
Keywords: COVID19; simvastatin; ruxolitinib
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — ruxolitinib; Simvastatin; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ruxolitinib plus simvastatin (Experimental): Ruxolitinib 5 mg orally every 12 hours for 7 days, which will be increased to 10 mg every 12 hours for a total of 14 days.
  Simvastatin 40 mg orally every 24 hours for 14 days.
  Interventions: Drug: Ruxolitinib plus simvastatin
- Standard of Care (Other): Patients will receive treatment according to usual clinical practice in the participant site.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: Ruxolitinib plus simvastatin — Ruxolitinib 5 mg orally every 12 hours for 7 days, which will be increased to 10 mg every 12 hours for a total of 14 days.
  Simvastatin 40 mg orally every 24 hours for 14 days
  Arms: Ruxolitinib plus simvastatin
Other: Standard of Care — Patients will receive treatment according to usual clinical practice in the participant site.
  Arms: Standard of Care

SUMMARY:
COVID-19's mechanism to enter the cell is initiated by its interaction with its cellular receptor, the angiotensin-converting enzyme. As a result of this union, a clathrin-mediated endocytosis process begins. This route is one of the therapeutic targets for which available drugs are being investigated in order to treat COVID-19 infection. This is one of the mechanisms blocked by drugs like ruxolitinib and chloroquine.

Various drugs approved for clinical use that block the clathrin-mediated endocytosis pathway have been explored. It has been found that the best in vitro and in vivo results were obtained with statins, which also allowed generating a greater potent adaptive immune response.

Therefore, statins and specifically simvastatin make it possible to block the entry process used by COVID-19, block inflammation by various mechanisms and increase the adaptive immune response. All of these processes are desirable in patients infected with COVID-19.

Statins have been proposed to have beneficial effects in patients infected with MERS-COV, another coronavirus similar to COVID-19, but there have been no randomized studies supporting the use of statins in patients with COVID-19 infection.

In this project we propose the combined use of one of these drugs, ruxolitinib with simvastatin, looking for a synergistic effect in the inhibition of viral entry and in the anti-inflammatory effect.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have given their written informed consent. If it is considered that obtaining written consent could constitute a factor for the transmission of the disease (given the high contagiousness of the SARS-Cov-2 virus), it will be permitted to obtain duly justified verbal consent in the patient's medical history.
* Clinical diagnosis or confirmed by analytical tests (PCR of viral RNA or detection of antiSARS-Cov-2 antibodies) that requires care in hospital and that are grade 3 or 4 of the WHO 7-point ordinal scale of severity categorization for COVID.
* Platelets> 50,000 / uL, neutrophils> 500 / ul
* Kidney or liver failure is not a contraindication, dose adjustment will be made according to the SmPC
* Women of childbearing potential who are sexually active, not undergoing a hysterectomy or double adnexectomy, should follow the following indications for contraception:

  * Negative serum or urine pregnancy test in the 72 hours prior to the start of treatment.
  * Use of a medically accepted contraceptive method during: 2 months prior to the start of study treatment, during the study and up to 3 months after the last dose of treatment.

Exclusion Criteria:

* Documented concomitant severe bacterial or fungal infection
* Infection with HIV, HCV, HBV
* Age <18 years
* Thrombocytopenia <50,000 / uL, Neutropenia <500 / uL
* Women of childbearing age who do not use an effective contraceptive method.
* Pregnant or lactating women.
* Patients who do not want or cannot comply with the protocol.
* Patients with impaired gastrointestinal function or gastric disease that significantly impairs the absorption of ruxolitinib or simvastatin, such as: severe ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, extensive resection (> 1m) of the small intestine or inability to swallow oral medication. Previous partial or total gastrectomy is not an exclusion criterion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2020-04-12 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who develop severe respiratory failure. | 7 days
  Patients achieving a grade 5 or higher of the WHO 7-point ordinal scale of severity categorization for COVID at day 7 from randomization.

SECONDARY OUTCOMES:
Percentage of patients who develop severe respiratory failure. | 14 days
  Patients achieving a grade 5 or higher of the WHO 7-point ordinal scale of severity categorization for COVID at day 14 from randomization.
Length of ICU stay. | 28 days
  Time from ICU admision to ICU discharge.
Length of hospital stay | 28 days
  Time from hospital admision to hospital discharge.
Survival rate at 6 months | 6 months
  Percentage of patients alive at 6 months
Survival rate at 12 months | 12 months
  Percentage of patients alive at 12 months
Survival rate at 28 days | 28 days
  Percentage of patients who died from any cause 28 days after inclusion in the study
Percentage of patients with each AE by grade | 28 days
  Percentage of patients with each AE by grade in relation with total number of treated patients
Percentage of patients who discontinued due to AEs | 28 days
  Percentage of patients who discontinued due to AEs in relation with total number of treated patients

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Madrid Sanchinarro, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Garcia-Donas J, Martinez-Urbistondo D, Velazquez Kennedy K, Villares P, Barquin A, Dominguez A, Rodriguez-Moreno JF, Caro E, Suarez Del Villar R, Nistal-Villan E, Yague M, Ortiz M, Barba M, Ruiz-Llorente S, Quiralte M, Zanin M, Rodriguez C, Navarro P, Berraondo P, Madurga R. Randomized phase II clinical trial of ruxolitinib plus simvastatin in COVID19 clinical outcome and cytokine evolution. Front Immunol. 2023 Apr 18;14:1156603. doi: 10.3389/fimmu.2023.1156603. eCollection 2023. PMID 37143685
- [Derived] Sultana J, Crisafulli S, Gabbay F, Lynn E, Shakir S, Trifiro G. Challenges for Drug Repurposing in the COVID-19 Pandemic Era. Front Pharmacol. 2020 Nov 6;11:588654. doi: 10.3389/fphar.2020.588654. eCollection 2020. PMID 33240091